CLINICAL TRIAL: NCT02718846
Title: A Multicenter, Randomized, Open-label Clinical Study With a Concurrent Control Group to Assess the Effectiveness and Safety of Combined Therapy With Isobide Solution and Meniace Tablets Compared to Monotherapy With Meniace Tablets for Patients With Meniere's Disease
Brief Title: Isobide Solution and Meniace Tablets Compared to Monotherapy With Meniace Tablets
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KW-ISOBIDE_P4
Record Dates: First submitted 2016-03-21; First posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Meniere's Disease
MeSH Terms: conditions — Meniere Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meniace and Isobide (Experimental): co-administration Isobide solution and Meniace tablets
  Interventions: Drug: Meniace; Drug: Isobide
- Meniace (Active Comparator): single administration Meniace tablets
  Interventions: Drug: Meniace

INTERVENTIONS:
Drug: Meniace — 6 mg of Meniace tablets were administered 3 times per day after meals
Drug: Isobide — an initial dosage of 90 mL of Isobide solution was administered orally 3 times a day after meals
  Arms: Meniace and Isobide

SUMMARY:
A multicenter, randomized, open-label clinical study with a concurrent control group to assess the effectiveness and safety of combined therapy with Isobide solution and Meniace tablets compared to monotherapy with Meniace tablets for patients with Meniere's disease

ELIGIBILITY:
Inclusion Criteria:

* 20 - 80 years of age (in full)
* A definite Meniere's disease patient according to the diagnostic criteria of AAO-HNS (1995), who has had 2 or more episodes of rotary dizziness lasting more than 20 minutes within the last 3 months (12 weeks) and 1 or more episodes of hearing loss recorded by audiometry, and has tinnitus or ear fullness.
* For female subjects with the possibility of pregnancy during the study period, a subject whose urine pregnancy test result was negative at the time of the screening visit. A subject in menopause for at least one year, one who has no possibility to become pregnant through surgery, or one who effectively uses an acceptable contraceptive measure. A subject who definitely agreed to use an adequate contraceptive measure during the clinical study period.

Exclusion Criteria:

* A patient with the history of ear surgery
* A patient with the history of endolymphatic sac surgery
* A patient who used steroids or gentamycin in the eardrum within the last 6 months
* A patient to whom Isobide was administered within 3 months at the time of screening
* A patient who has an infection in the ear, paranasal sinuses or the upper airway system
* A patient who has a disease, other than Meniere's disease, that manifests as repetitive dizziness (e.g. Migrainous vertigo, vertebrobasilar transient ischemic attack, acoustic neuroma)
* A patient who has acute intracranial hematoma (If this drug is administered to a patient suspected of having an acute intracranial hematoma without checking for the existence of an intracranial hematoma, bleeding that had been stopped temporarily by brain pressure can occur again when intracranial pressure is reduced. Thus, eliminate the cause of bleeding and administer the drug after ensuring that there are no concerns of rebleeding)
* A patient with anuria (with urinary output of less than 100 mL/day)
* A severely dehydrated patient (loss of 10% or more of body weight)
* A patient with acute pulmonary edema
* A patient with severe heart failure (New York Heart Association class III or higher)
* A patient with an adrenal tumor
* A patient with pheochromocytoma
* A patient who is hypersensitive to the ingredients of the test and control drugs
* A patient with a hereditary disease such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption
* A woman who is pregnant or breastfeeding
* A patient who is deemed ineligible for this clinical study by the analyst

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2013-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
the number of vertigo episodes | The difference between the number of vertigo episodes experienced during the 4 weeks before the screening and the number of vertigo episodes during the 4 weeks after administration of the study drug

CONTACTS AND LOCATIONS:
Overall Officials: Won-ho Jeong, Ph.D., Principal Investigator — Samsung Medical Center

IPD SHARING:
Plan to Share IPD: No